CLINICAL TRIAL: NCT02908789
Title: Evaluation of Antimicrobial Photodynamic Therapy as an Adjunct Treatment for Deep Carious Lesions in Children
Brief Title: Evaluation of Antimicrobial Photodynamic Therapy as an Adjunct Treatment of Deep Carious Lesions in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Livia Azeredo Alves Antunes, Professor Lívia Azeredo Alves Antunes, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PDTa and dental carie
Record Dates: First submitted 2016-09-01; First posted 2016-09-21 (Estimated); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Dental Caries
Keywords: Photochemotherapy
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Antimicrobial photodynamic therapy (aPDT) (Experimental): 1)Selective caries removal: caries dentin was partially removed with hand excavators (Fava, Pirituba, Brazil). 2)The laser technique: 0.01% methylene blue solution was applied, and a pre-irradiation period of 5 minutes was done with an Indium Gallium Aluminum Phosphorus diode laser (InGaAlP) with a wavelength of 660 nm (visible red), a spot area of 3mm2, and fixed output power of 100 mW (energy of 9 J with 90 seconds). 3) The restorative technique was done as described in comparator group.
  Interventions: Radiation: Antimicrobial photodynamic therapy (aPDT)
- Group without Antimicrobial photodynamic therapy (aPDT) (Sham Comparator): 1) Selective caries removal 2) The restorative technique was done by etching with 37% CondacTM phosphoric acid conditioner (FGM) for 15 s in enamel and 7 s in dentin was performed followed by washing for 30 s until the conditioner was completely removed. The excess of dentin moisture was removed with sterile cotton balls, and the enamel was air-dried until it had an opaque appearance. Subsequently, two consecutive layers of Adper Single Bond 2TM (3M ESPE) were applied with a KG Brush (KG Sorensen) on the enamel and dentin for 15 s and subjected to light air blast to promote solvent evaporation. The adhesive was photoactivated for 10 s with a light-emitting diode (LED) unit (BioLuz Plus; BioArt) with an intensity of 460 mW/mm2. The cavity was restored with a Filtek Z250TM composite resin (3M Dental Products) according to the incremental technique. Each increment was photo-activated for 40 s.
  Interventions: Other: Without Antimicrobial phothodynamic therapy

INTERVENTIONS:
Radiation: Antimicrobial photodynamic therapy (aPDT) — Selective caries removal + Antimicrobial photodynamic therapy (aPDT) is an effective low potency laser that involves the activation of a photosensitizer( 0.01% methylene blue ) by a visible light source that creates chemical reactions, producing cytotoxic reactive oxygen species and causing oxidative stress and inactivation of pathogenic microorganisms + tooth restauration
  Arms: Antimicrobial photodynamic therapy (aPDT)
Other: Without Antimicrobial phothodynamic therapy — Selective caries removal + tooth restauration
  Arms: Group without Antimicrobial photodynamic therapy (aPDT)

SUMMARY:
This project aims to evaluate the effect of antimicrobial photodynamic therapy (aPDT) in deep carious lesions. This study was approved by the Research Ethics Committee and was conducted on 53 patients between 3 and 12 years. Patients included in the study should have at least one primary molar or permanent with deep active caries and limited occlusal/proximal surfaces involving beyond the inner half of dentin. The investigators considered from exclusion criteria children whose parents refuse to sign the informed consent document; children who do not cooperate with the clinical examination/treatment; children with syndromes or chronic systemic diseases; teeth with painful symptoms consistent with irreversible pulpitis or mobility; periodontal changes; roots with pathological resorption; cases of primary teeth roots in an advanced stage of physiological resorption and patients that have made the use of any antibiotics during the study period or within three months prior to its beginning. The treatments were carried out after local anesthesia and isolation of the operative field with a rubber dam. The removal of carious dentin surface demineralized necrotic and not subject to remineralization was held with the drill at low rpm under cooling with sterile saline. The removal of decayed tissue will start with the side walls and later on the pulp wall. After this time the intervention with aPDT using 0.01% methylene blue as photosensitizer will be held. Finally, the cavity is restored with an adhesive and composite resin system. To collect data for the first outcome the dentin samples were collected from 23 participants with the help of spoon sterile dentine in two stages: C1 after digging and C2 after aPDT. The microbiological analyzes will be conducted by counting colony-forming units (CFU / mg of carious dentin), blindly from coded samples. The viability of microorganisms will be evaluated in the following culture media: Brain Heart Infusion agar for the feasibility of total microorganisms; CHROMagar candida to Candida genus; Mitis Salaviarius agar with the addition of bacitracin 0.2 U/mL, sucrose and glucose to Streptococcus mutans; Mitis Salivarius agar to total Streptococcus; Rogosa Agar to Lactobacillus spp. and enterococcosel for Enterococcus genus. The reproducibility of the counting method will be verified between triplicates. Microbiological data will be evaluated with appropriate statistical tests with a level of 5%. For the second outcome, a randomized clinical trial was designed. Primary molars of 30 patients (mean age 6.15 years) with deep caries lesions without signs and symptoms of pulpal involvement were selected. A total of 64 teeth were randomly divided into groups G1 (SCR, 32 teeth) and G2 (SCR + aPDT, 32 teeth) for treatment, restored with composite and evaluated after a week (T0), 6 months (T1), and 12 months (T2) according to the criteria of FDI. Groups were compared using the Rao-Scott chi-squared test and the logistic regression analysis for complex designs to ac- count for multiple observations per subject (alpha = 0.05). All participants answered a questionaire to detect the impact on Oral Health-related quality of life(OHRQoL) before and 3 months after the treatment. Based on this project we prove the clinical efficacy of aPDT using 0.01% methylene blue as an adjunct in reducing microorganisms from the interior of deep carious lesions and we contributed to demonstrate the clinical and radiographic success in a follow-up from 12 months providing additional support aPDT used as an adjunct to SCR on the longevity of composite resin restorations in primary molars. A low laser therapy (aPDT) with SCR did not influence negatively OHRQoL. In the practice of pediatric dentistry, this conservative dental treatment improved the OHRQoL after 3 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study should have at least one primary molar or permanent with deep active caries limited occlusal / proximal surfaces involving beyond the inner half of dentin.

Exclusion Criteria:

* Children whose parents refuse to sign the informed consent document
* Children who do not cooperate with the clinical examination/treatment
* Children with syndromes or chronic systemic diseases
* Teeth with painful symptoms consistent with irreversible pulpitis or mobility
* Periodontal changes
* Roots with pathological resorption
* Cases of primary teeth roots in advanced stage of physiological resorption and patients that have made the use of any antibiotics during the study period or within three months prior to its beginning

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Evaluate Antimicrobial photodynamic therapy (aPDT) on microorganism reduction in deep cavities immediately after dental caries remotion and immediately use aPDT | Microorganisms reduction couting of colony forming units will be evaluated seven days after. The clinical success will be evaluated 3 months, 6 months, 12 months and 24 months.
  Microorganisms reduction count after after manual excavation (control) and immediately after aPDT (experimental) obtained by means counting of colony forming units (CFU / mg of carious dentin), blindly from coded samples from the following viability of microorganisms total microorganisms; Candida genus; Streptococcus mutans; total Streptococcus; Lactobacillus spp. and for Enterococcus genus.After the period of 3, 6, 12 and 24 months of implementation of the treatment, there will be clinical and radiographic examination for treatment success.
Evaluation of composite restorations in primary molars subjected to selective caries removal associated with antimicrobial photodynamic therapy | A total of 64 teeth were randomly divided into groups G1 (SCR, 32 teeth) and G2 (SCR + aPDT, 32 teeth) for treatment, restored with composite, and evaluated after a week (T0), 6 months (T1), and 12 months (T2) according to the criteria of FDI.
  Antimicrobial photodynamic therapy (aPDT) has been used as an adjunct treatment of deep caries lesions; however, studies on the effects of aPDT on the longevity of restorations are still limited.

SECONDARY OUTCOMES:
Effect of Treatment with Selective Caries Removal Associated to Antimicrobial Photodynamic Therapy on Children's Oral HealthRelated Quality of Life: A Non-Randomized Clinical Study | The impact was assessed before and after conservative treatment of deep caries lesions using the selective caries removal (SCR) associated to a low laser therapy (antimicrobial photodynamic therapy-aPDT) on oral health-related quality of life (OHRQoL).
  How patients perceive impact of diseases is an essential component when characterising different disease impacts, and effects of dental treatments should be perceived by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Livia Antunes, PHD, Principal Investigator — Universidade Federal Fluminense
Locations (1):
- Universidade Federal Fluminense, Nova Friburgo, Rio de Janeiro, Brazil